CLINICAL TRIAL: NCT04636255
Title: Physical Capacity Evaluation and Effects of ExerciseTraining on Hodgkin Lymphoma Survivors
Brief Title: Physical Capacity in Hodgkin Lymphoma Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 432715154
Record Dates: First submitted 2020-11-12; First posted 2020-11-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-05

CONDITIONS: Hodgkin Lymphoma, Adult; Cardiovascular Diseases; Radiation Effect; Chemotherapy Effect
Keywords: Oxygen Consumption; Physical Training; Heart Hate; Cardioprotection
MeSH Terms: conditions — Hodgkin Disease; Cardiovascular Diseases | interventions — Blood Pressure; Physical Conditioning, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training group (Experimental): Patients in the experimental group, under clinic follow up will perform combined exercise training for 16 weeks
  Interventions: Procedure: Physical Characteristics; Diagnostic Test: Assessment of Heart rate variability; Diagnostic Test: Blood Pressure and Cardiac Autonomic Control; Diagnostic Test: Evaluation of Baroreflex Control; Diagnostic Test: Cardiac Function and Structure; Diagnostic Test: Assessment of Coronary Anatomy and Calcium Score; Diagnostic Test: Blood Assessments; Diagnostic Test: Physical Capacity; Procedure: Physical Training
- Control Group (Sham Comparator): Patients will be only clinically followed up. They will not perform exercise training.
  Interventions: Procedure: Physical Characteristics; Diagnostic Test: Assessment of Heart rate variability; Diagnostic Test: Blood Pressure and Cardiac Autonomic Control; Diagnostic Test: Evaluation of Baroreflex Control; Diagnostic Test: Cardiac Function and Structure; Diagnostic Test: Assessment of Coronary Anatomy and Calcium Score; Diagnostic Test: Blood Assessments; Diagnostic Test: Physical Capacity

INTERVENTIONS:
Procedure: Physical Characteristics — Body Weight, Height
Diagnostic Test: Assessment of Heart rate variability — Holter 24h
Diagnostic Test: Blood Pressure and Cardiac Autonomic Control — Non-invasive photoplethysmography (Finometer® PRO) monitored by the electrocardiogram and respiratory frequency by a piezoelectric chest strap.
Diagnostic Test: Evaluation of Baroreflex Control — The magnitude and latency of the baroreflex control of the heart rate will be assessed by bivariate analysis using the autoregressive method.
Diagnostic Test: Cardiac Function and Structure — Echocardiogram
Diagnostic Test: Assessment of Coronary Anatomy and Calcium Score — Angiotomography
Diagnostic Test: Blood Assessments — Serum and Plasma will be extracted by centrifugation. NT-pro BNP (Roche™) and c-TnI (imunoassay Elecys 2010).
Diagnostic Test: Physical Capacity — Cardiopulmonary Exercise Test.
Procedure: Physical Training — Aerobic exercise: 48 sessions of 60 minutes: 5 minutes of warm-up, 40 minutes of exercise. Resistance exercise: 10 minutes of exercise and 5 minutes of recovery.
  Arms: Exercise training group

SUMMARY:
The study aims to investigate if physical capacity obtained in the cardiopulmonary exercise test can predict cardiovascular alterations in Hodgkin Lymphoma (HL) Survivors. In addition, to study the effects of exercise training on physical capacity and cardiovascular responses in these patients.

DETAILED DESCRIPTION:
Hodgkin Lymphoma (HL) is a hematological neoplasia that mainly affects young people. Anthracycline-based chemotherapy, followed or not by mediastinal radiotherapy, substantially improves prognosis in this set of patients. Observational studies have shown that cardiovascular disease is the most non oncologic cause of death in this population. Coronary artery disease (CAD) affects 26% of survivors after 10 years of absence of HL . However, the early intervention and the assessment to predict the cardiovascular risk remain little known. In this study, the investigators will test the hypothesis that physical capacity can predict the cardiovascular alterations in HL Survivors. In addition, exercise training improves physical capacity and heart rate responses in this set of patients.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin Lymphoma Survivors
* Over 18 years old
* Chemotherapy with anthracycline and mediastinal radiotherapy in the last 5 years or more

Exclusion Criteria:

* Renal insufficiency
* Pregnant women,
* Iodinated contrast allergy,
* Life expectancy less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10-21 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2023-10-21 (Estimated)

PRIMARY OUTCOMES:
Physical Capacity - Peak oxygen consumption (mL/kg/min) | 4 months
  Oxygen consuption in crescent effort will be calculated by aggregation of volume (mL), body weight (Kg) and time (minutes).

SECONDARY OUTCOMES:
Heart Hate (beat/min) | 4 months
  Post-exercise heart rate will be evaluated by the number of beats in time masurement (one minute).
Cardiac Function - Ejection Fraction | 4 months
  Ejection Fraction (EF=ESV-EDV/EDV) combines end systolic (ESV) and diastolic volumes (EDV)(mL)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Negrao, PhD, Principal Investigator — Instituto do Coracao, HCFMUSP, Faculdade de Medicina, Universidade de Sao Paulo
Locations (1):
- Luciana de Souza Santos, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ansell SM. Hodgkin Lymphoma: Diagnosis and Treatment. Mayo Clin Proc. 2015 Nov;90(11):1574-83. doi: 10.1016/j.mayocp.2015.07.005. PMID 26541251
- [Background] Heidenreich PA, Schnittger I, Strauss HW, Vagelos RH, Lee BK, Mariscal CS, Tate DJ, Horning SJ, Hoppe RT, Hancock SL. Screening for coronary artery disease after mediastinal irradiation for Hodgkin's disease. J Clin Oncol. 2007 Jan 1;25(1):43-9. doi: 10.1200/JCO.2006.07.0805. PMID 17194904
- [Background] Gilchrist SC, Barac A, Ades PA, Alfano CM, Franklin BA, Jones LW, La Gerche A, Ligibel JA, Lopez G, Madan K, Oeffinger KC, Salamone J, Scott JM, Squires RW, Thomas RJ, Treat-Jacobson DJ, Wright JS; American Heart Association Exercise, Cardiac Rehabilitation, and Secondary Prevention Committee of the Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; and Council on Peripheral Vascular Disease. Cardio-Oncology Rehabilitation to Manage Cardiovascular Outcomes in Cancer Patients and Survivors: A Scientific Statement From the American Heart Association. Circulation. 2019 May 21;139(21):e997-e1012. doi: 10.1161/CIR.0000000000000679. PMID 30955352
- [Background] Girinsky T, M'Kacher R, Lessard N, Koscielny S, Elfassy E, Raoux F, Carde P, Santos MD, Margainaud JP, Sabatier L, Ghalibafian M, Paul JF. Prospective coronary heart disease screening in asymptomatic Hodgkin lymphoma patients using coronary computed tomography angiography: results and risk factor analysis. Int J Radiat Oncol Biol Phys. 2014 May 1;89(1):59-66. doi: 10.1016/j.ijrobp.2014.01.021. Epub 2014 Mar 7. PMID 24613809
- [Background] Hoppe RT, Advani RH, Ai WZ, Ambinder RF, Aoun P, Bello CM, Bierman PJ, Blum KA, Chen R, Dabaja B, Duron Y, Forero A, Gordon LI, Hernandez-Ilizaliturri FJ, Hochberg EP, Maloney DG, Mansur D, Mauch PM, Metzger M, Moore JO, Morgan D, Moskowitz CH, Poppe M, Pro B, Winter JN, Yahalom J, Sundar H; National Comprehensive Cancer Network. Hodgkin lymphoma, version 2.2012 featured updates to the NCCN guidelines. J Natl Compr Canc Netw. 2012 May;10(5):589-97. doi: 10.6004/jnccn.2012.0061. PMID 22570290
- [Background] Kavanagh T, Mertens DJ, Hamm LF, Beyene J, Kennedy J, Corey P, Shephard RJ. Prediction of long-term prognosis in 12 169 men referred for cardiac rehabilitation. Circulation. 2002 Aug 6;106(6):666-71. doi: 10.1161/01.cir.0000024413.15949.ed. PMID 12163425
- [Background] Aleman BM, van den Belt-Dusebout AW, De Bruin ML, van 't Veer MB, Baaijens MH, de Boer JP, Hart AA, Klokman WJ, Kuenen MA, Ouwens GM, Bartelink H, van Leeuwen FE. Late cardiotoxicity after treatment for Hodgkin lymphoma. Blood. 2007 Mar 1;109(5):1878-86. doi: 10.1182/blood-2006-07-034405. Epub 2006 Nov 21. PMID 17119114
- [Background] Koelwyn GJ, Jones LW, Moslehi J. Unravelling the causes of reduced peak oxygen consumption in patients with cancer: complex, timely, and necessary. J Am Coll Cardiol. 2014 Sep 30;64(13):1320-2. doi: 10.1016/j.jacc.2014.07.949. No abstract available. PMID 25257632
- [Background] Groarke JD, Tanguturi VK, Hainer J, Klein J, Moslehi JJ, Ng A, Forman DE, Di Carli MF, Nohria A. Abnormal exercise response in long-term survivors of hodgkin lymphoma treated with thoracic irradiation: evidence of cardiac autonomic dysfunction and impact on outcomes. J Am Coll Cardiol. 2015 Feb 17;65(6):573-83. doi: 10.1016/j.jacc.2014.11.035. PMID 25677317
- [Background] Wilson MG, Ellison GM, Cable NT. Basic science behind the cardiovascular benefits of exercise. Heart. 2015 May 15;101(10):758-65. doi: 10.1136/heartjnl-2014-306596. PMID 25911667
- [Background] da Silva VP, de Oliveira NA, Silveira H, Mello RG, Deslandes AC. Heart rate variability indexes as a marker of chronic adaptation in athletes: a systematic review. Ann Noninvasive Electrocardiol. 2015 Mar;20(2):108-18. doi: 10.1111/anec.12237. Epub 2014 Nov 26. PMID 25424360
- [Background] Cramer L, Hildebrandt B, Kung T, Wichmann K, Springer J, Doehner W, Sandek A, Valentova M, Stojakovic T, Scharnagl H, Riess H, Anker SD, von Haehling S. Cardiovascular function and predictors of exercise capacity in patients with colorectal cancer. J Am Coll Cardiol. 2014 Sep 30;64(13):1310-9. doi: 10.1016/j.jacc.2014.07.948. PMID 25257631
- [Background] Pumprla J, Howorka K, Groves D, Chester M, Nolan J. Functional assessment of heart rate variability: physiological basis and practical applications. Int J Cardiol. 2002 Jul;84(1):1-14. doi: 10.1016/s0167-5273(02)00057-8. PMID 12104056